CLINICAL TRIAL: NCT01326650
Title: Effect of Vitamin D on All-cause Mortality in Heart Failure Patients
Brief Title: Vitamin D and Mortality in Heart Failure
Acronym: EVITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2015-09

CONDITIONS: Congestive Heart Failure
Keywords: vitamin D, mortality, event-free survival, heart failure
MeSH Terms: conditions — Heart Failure | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Experimental): daily vitamin D supplement
  Interventions: Drug: Vitamin D
- placebo (Placebo Comparator): daily placebo supplement
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D — daily oral vitamin D supplement of 100 micrograms for three years
  Other Names: solution of vitamin D oil
  Arms: Vitamin D
Drug: placebo — daily oral placebo supplement for three years
  Other Names: solution of migliol oil
  Arms: placebo

SUMMARY:
Despite significant therapeutic improvements, congestive heart failure (CHF) patients still have a poor prognosis. Currently, 5-year survival rates are only 35-50%. There is an accumulating body of evidence from prospective cohort studies that low circulating 25-hydroxyvitamin D is an independent predictor of all-cause and cardiovascular mortality, respectively. Vitamin D deficiency is prevalent among CHF patients. We hypothesize that vitamin D may improve survival in CHF patients. We therefore aimed to investigate whether vitamin D supplementation reduces mortality and increases event-free survival in end-stage CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age and < 80 years of age
* New York Heart Association Functional Class > = II

Exclusion Criteria:

* pregnancy and lactation
* sarcoidosis
* daily vitamin D intake > 20 micrograms
* serum 25-hydroxyvitamin D > 30 ng/ml
* hypercalcemia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who died during the intervention | three years
  all-cause mortality (any cause of death) will be assessed

SECONDARY OUTCOMES:
Number of event-free survivors | three years
  event defined as: cardiac transplantation, high urgent listing for cardiac transplantation, resuscitation, ventricular assist device Implantation, hypercalcemia
Changes in biochemical risk markers | three years
  inflammation markers, kidney parameters, lipid parameters, haemostasis parameters
Number of participants with elevated safety parameters | every 6 months
  Serum 25-Hydroxyvitamin D should not exceed 150 ng/ml.
  Serum calcium should not exceed 2.75 mmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Zittermann, PhD, Study Chair — Heart Center North Rhine-Westphalia; Jochen Börgermann, MD, Principal Investigator — Heart Center North Rhine-Westphalia
Locations (1):
- Heart Center North Rhine-Westphalia, Bad Oeynhausen, Federal State of North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Zittermann A, Schleithoff SS, Frisch S, Gotting C, Kuhn J, Koertke H, Kleesiek K, Tenderich G, Koerfer R. Circulating calcitriol concentrations and total mortality. Clin Chem. 2009 Jun;55(6):1163-70. doi: 10.1373/clinchem.2008.120006. Epub 2009 Apr 9. PMID 19359534
- [Background] Zittermann A, Frisch S, Berthold HK, Gotting C, Kuhn J, Kleesiek K, Stehle P, Koertke H, Koerfer R. Vitamin D supplementation enhances the beneficial effects of weight loss on cardiovascular disease risk markers. Am J Clin Nutr. 2009 May;89(5):1321-7. doi: 10.3945/ajcn.2008.27004. Epub 2009 Mar 25. PMID 19321573
- [Background] Zittermann A, Schleithoff SS, Gotting C, Fuchs U, Kuhn J, Kleesiek K, Tenderich G, Koerfer R. Calcitriol deficiency and 1-year mortality in cardiac transplant recipients. Transplantation. 2009 Jan 15;87(1):118-24. doi: 10.1097/TP.0b013e31818c2708. PMID 19136901
- [Background] Zittermann A, Schleithoff SS, Gotting C, Dronow O, Fuchs U, Kuhn J, Kleesiek K, Tenderich G, Koerfer R. Poor outcome in end-stage heart failure patients with low circulating calcitriol levels. Eur J Heart Fail. 2008 Mar;10(3):321-7. doi: 10.1016/j.ejheart.2008.01.013. Epub 2008 Mar 4. PMID 18304873
- [Background] Zittermann A, Fischer J, Schleithoff SS, Tenderich G, Fuchs U, Koerfer R. Patients with congestive heart failure and healthy controls differ in vitamin D-associated lifestyle factors. Int J Vitam Nutr Res. 2007 Jul;77(4):280-8. doi: 10.1024/0300-9831.77.4.280. PMID 18271283
- [Background] Schleithoff SS, Zittermann A, Tenderich G, Berthold HK, Stehle P, Koerfer R. Vitamin D supplementation improves cytokine profiles in patients with congestive heart failure: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2006 Apr;83(4):754-9. doi: 10.1093/ajcn/83.4.754. PMID 16600924
- [Background] Zittermann A, Schleithoff SS, Tenderich G, Berthold HK, Korfer R, Stehle P. Low vitamin D status: a contributing factor in the pathogenesis of congestive heart failure? J Am Coll Cardiol. 2003 Jan 1;41(1):105-12. doi: 10.1016/s0735-1097(02)02624-4. PMID 12570952
- [Derived] Zittermann A, Ernst JB, Prokop S, Fuchs U, Dreier J, Kuhn J, Knabbe C, Borgermann J, Berthold HK, Pilz S, Gouni-Berthold I, Gummert JF. Daily Supplementation with 4000 IU Vitamin D3 for Three Years Does Not Modify Cardiovascular Risk Markers in Patients with Advanced Heart Failure: The Effect of Vitamin D on Mortality in Heart Failure Trial. Ann Nutr Metab. 2019;74(1):62-68. doi: 10.1159/000495662. Epub 2018 Dec 14. PMID 30554193
- [Derived] Ernst JB, Prokop S, Fuchs U, Dreier J, Kuhn J, Knabbe C, Berthold HK, Pilz S, Gouni-Berthold I, Gummert JF, Borgermann J, Zittermann A. Randomized supplementation of 4000 IU vitamin D3 daily vs placebo on the prevalence of anemia in advanced heart failure: the EVITA trial. Nutr J. 2017 Aug 23;16(1):49. doi: 10.1186/s12937-017-0270-5. PMID 28835271
- [Derived] Zittermann A, Ernst JB, Prokop S, Fuchs U, Dreier J, Kuhn J, Knabbe C, Birschmann I, Schulz U, Berthold HK, Pilz S, Gouni-Berthold I, Gummert JF, Dittrich M, Borgermann J. Effect of vitamin D on all-cause mortality in heart failure (EVITA): a 3-year randomized clinical trial with 4000 IU vitamin D daily. Eur Heart J. 2017 Aug 1;38(29):2279-2286. doi: 10.1093/eurheartj/ehx235. PMID 28498942